CLINICAL TRIAL: NCT01402193
Title: A Prospective, Randomized, Bi-center Study to Compare the Outcome of Adjuvant Radiotherapy With Concomitant or Sequential Arimidex in Postmenopausal Women With Breast Cancer
Brief Title: Study of Arimidex and Radiotherapy Sequencing
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Jiayi Chen, Associate Professor, Vice Chairman of Department of Radiation Oncology, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BR-RT-002
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Timing of Radiotherapy; TGF-beta1
MeSH Terms: conditions — Breast Neoplasms; Camurati-Engelmann Syndrome | interventions — Anastrozole; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Arm (Active Comparator): Investigational treatment: Arimidex commenced before and continued during radiotherapy.
  Interventions:
  Drug: Pre-radiotherapy commencement of Arimidex Radiation: Radiotherapy
  Interventions: Drug: Pre-radiotherapy commencement of Arimidex; Radiation: Radiotherapy
- Control Arm (Active Comparator): Standard Treatment: Arimidex delayed until 2 weeks after radiotherapy
  Interventions:
  Radiation: Radiotherapy Drug: Post radiotherapy commencement of Arimidex
  Interventions: Drug: Post radiotherapy commencement of Arimidex; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Pre-radiotherapy commencement of Arimidex — Arimidex:1mg P.O. daily will be prescribed for 8 weeks in post-mastectomy patients and 9 weeks in BCT patients within the study period. Arimidex starts 3 weeks before adjuvant radiotherapy and throughout the course of radiotherapy.Total duration of adjuvant hormonotherapy is prescribed by the investigators at the completion of study, 5 years in principle.
  Other Names: Anastrozole
  Arms: Study Arm
Drug: Post radiotherapy commencement of Arimidex — Arimidex：1mg P.O. daily will be prescribed at 2 weeks after the end of radiotherapy.Total duration of adjuvant hormonotherapy is prescribed by the investigators at the completion of study, 5 years in principle.
  Other Names: Anastrozole
  Arms: Control Arm
Radiation: Radiotherapy — Radiotherapy is delivered to the whole breast/chest wall +/- regional lymph nodes to a total dose of 50Gy/25 fractions/5weeks, an additional tumor bed boost of 10Gy/5 fractions/1week is delivered to patients with breast conservative surgery
  Other Names: RT, Radiation Therapy
  Arms: Study Arm
Radiation: Radiotherapy — Radiotherapy is delivered to the whole breast/chest wall +/- regional lymph nodes to a total dose of 50Gy/25 fractions/5weeks, an additional tumor bed boost of 10Gy/5 fractions/1week is delivered to patients with breast conservative surgery
  Other Names: RT, Radiation Therapy
  Arms: Control Arm

SUMMARY:
The purpose of this study is to compare TGF-β1 change in concomitant with that in sequential Arimidex in postmenopausal women with breast cancer, as measured by the proportion of patients with an elevation of TGF-β1 level at the 4th week after initiation of radiotherapy relative to the pre-treatment baseline.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Pathological confirmation of breast cancer
* ER(+) and/or PR(+).
* Post-menopausal woman
* Age≤70 years old
* Breast conservative surgery with axillary dissection or staging by either sentinel nodes biopsy or axillary sampling
* Post-mastectomy patients with T1-T2 and N1-N3, or T3-T4 with any N Negative surgical margins
* Karnofsky≥70
* Laboratory criteria:

  * PLT≥100*109/L
  * WBC≥4000/mm3
  * HGB≥10g/dl
  * ALT and AST<2*ULN
* No presence of metastatic disease
* No other malignant tumour

Exclusion Criteria:

* Presence of metastatic disease.
* T1, T2, N0 with mastectomy
* Non-infiltrative breast carcinoma underwent mastectomy
* Other malignant tumor (concurrent or previous).
* Positive surgical margins.
* Patients with demonstrated hypersensitivity to Arimidex or any excipient.
* Patients with severe renal impairment (creatinine clearance less than 20 ml/min).
* Patients with moderate or severe hepatic disease.
* Oestrogen-containing therapies should not be co-administered with Arimidex as they would negate its pharmacological action.
* Not able or willing to sign informed consent
* Autoimmune diseases including scleroderma, systemic lupus erythematosus and so on

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-12 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Level of TGF-β1 | First analysis will occur 1 year after first subject enrolled
  To compare TGF-β1 change in concomitant with that in sequential Arimidex in postmenopausal women with breast cancer, as measured by the proportion of patients with an elevation of TGF-β1 level at the 4th week after initiation of radiotherapy relative to the pre-treatment baseline.

SECONDARY OUTCOMES:
Acute skin reaction | First analysis will occur 1 year after first subject enrolled
  Acute skin reaction occurrence rate defined by the occurrence of grade II or above acute skin reaction in patients with concurrent or sequential arimidex with radiotherapy.
Other serum inflammatory cytokine | First analysis will occur 1 year after first subject enrolled
  Pre-and post-radiotherapy other serum inflammatory cytokine
Cosmetic outcomes | First analysis will occur 1 year after first subject enrolled
  Cosmetic outcomes in patients receiving breast conservative therapy treated by both arms.
Lung toxicity | First analysis will occur 1 year after first subject enrolled
  Occurrence of grade II or higher radiation-induced lung toxicity.
Local-regional recurrence | First analysis will occur 1 year after first subject enrolled
  Local-regional recurrence within two arms.
Correlation between TGF-β1 Change and Clinical Outcomes | First analysis will occur 1 year after first subject enrolled
  The correlation between TGF-β1 change and clinical outcomes will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayi Chen, MD, Principal Investigator — The Department of Radiation Oncology, Fudan University Cancer Hospital
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China